CLINICAL TRIAL: NCT06637488
Title: Correction of Cleft Nasal Deformity Using Customized Milled Nasal Conformer in Unilateral Cleft Lip Repair (a Randomized Controlled Clinical Trial )
Brief Title: Using Customized Nasal Conformer in Correction of Cleft Nasal Deformity in Patients with Unilateral Cleft Lip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Akram (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Akram, Assistant lecturer of Oral and Maxillofacial surgery, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nasal conformer in cleft lip
Record Dates: First submitted 2024-10-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Unilateral Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unilateral cleft lip repair using customized nasal conformer (Experimental)
  Interventions: Procedure: cleft lip repair using fisher technique
- Unilateral cleft lip repair without using customized nasal conformer (Active Comparator)
  Interventions: Procedure: cleft lip repair using fisher technique

INTERVENTIONS:
Procedure: cleft lip repair using fisher technique — Disinfection of the field using Betadine , marking for the incision lines on the lip and vermilion on skin and mucosa , doing incisions as described by Fisher sub anatomic unit repair in 2005 , suturing using vicryl and prolene sutures. suturing the nasal conformer in the cleft side
  Arms: Unilateral cleft lip repair using customized nasal conformer
Procedure: cleft lip repair using fisher technique — Disinfection of the field using Betadine , marking for the incision lines on the lip and vermilion on skin and mucosa , doing incisions as described by Fisher sub anatomic unit repair in 2005 , suturing using vicryl and prolene sutures. No nasal conformers used in this group
  Arms: Unilateral cleft lip repair without using customized nasal conformer

SUMMARY:
The goal of the study is to compare the cleft lip repair with and without the usage of customized milled nasal conformers in unilateral cleft lip patients on nostril size , alar cartilage and proportion of symmetry to the normal side .

* Comparing anthropometric measurements similarity between cleft and normal sides such as; nostril width and height , columellar deviation and nasolabial angle.
* Evaluation of degree of similarity using esthetic scales at six months postoperative.

Participants will receive nasal conformers intraoperative with follow up of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes with unilateral cleft lip.
2. Age range 10 - 24 weeks.
3. Hemoglobin more than 10 gm/dl .
4. Weight more than 10 lbs.

Exclusion Criteria:

1. Syndromic patients.
2. Patients with conditions contradicting operation.
3. Patients with Bilateral cleft lip.
4. Patients with previous surgeries in lip and nose.

Ages: 10 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Nostril height | 6 months
  The greatest vertical distance of the nostril in millimeters .
Nostril width | 6 months
  This measure was defined as the greatest horizontal distance between the inner medial and lateral borders of the nostril aperture in millimeters.
Columellar Deviation Angle | 6 months
  The midline columellar deviation from the vertical reference line was measured in degrees.
Nasolabial Groove Angle | 6 months
  To assess the flare of the nasal alar base, the angle between a line tangential to the outer alar basepoint and the horizontal reference line was measured in degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khodir MA, Osman SM, Ragab HR, AboulHassan MA, Oraby MS. Assessment of symmetry and parental satisfaction after use of customized nasal conformers in unilateral cleft lip repair: a randomized controlled clinical trial. Head Face Med. 2025 Aug 1;21(1):55. doi: 10.1186/s13005-025-00533-6. PMID 40751267